CLINICAL TRIAL: NCT02530190
Title: Investigation of Popular Recovery Techniques for Ultramarathon Recovery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Western States Endurance Run Research Foundation (Other)
Responsible Party: Principal Investigator, Martin D. Hoffman, MD, Director of Research, Western States Endurance Run Research Foundation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WSER 2015
Record Dates: First submitted 2015-08-18; First posted 2015-08-20 (Estimated); Last update posted 2015-08-20 (Estimated); Status verified 2015-08

CONDITIONS: Musculoskeletal Pain
MeSH Terms: conditions — Musculoskeletal Pain | interventions — Intermittent Pneumatic Compression Devices; Massage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (No Intervention): 20 minutes of supine rest
- Intermittent pneumatic compression (Active Comparator): 20 minutes of intermittent pneumatic compression
  Interventions: Device: intermittent pneumatic compression
- Massage (Active Comparator): 20 minutes of massage therapy
  Interventions: Procedure: massage

INTERVENTIONS:
Device: intermittent pneumatic compression — 20 minutes of intermittent pneumatic compression to lower extremities
  Arms: Intermittent pneumatic compression
Procedure: massage — 20 minutes of massage to lower extremities
  Arms: Massage

SUMMARY:
The study is a randomized clinical trial examining the effectiveness of massage and intermittent pneumatic compression on recovery from a 161-km ultramarathon.

DETAILED DESCRIPTION:
The study is a randomized clinical trial examining the effectiveness of massage and intermittent pneumatic compression on recovery from a 161-km ultramarathon. Participants of the 2015 161-km Western States Endurance Run were randomized to a 20-minute post-race intervention of massage, intermittent pneumatic compression or supine rest. Each subject completed two 400 m runs at maximum speed before the race, and on days 3 and 5 after the race, and also provided muscle pain and soreness ratings and overall muscular fatigue scores before and for 7 days after the race.

ELIGIBILITY:
Inclusion Criteria:

* Entry in the Western States Endurance Run

Exclusion Criteria:

* Failure to finish race

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2015-05; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
400 m run time | 5 days
  self-timed 400 m run as fast as possible

SECONDARY OUTCOMES:
Lower body muscle pain and soreness rating | 5 days
  Subjective rating of lower body muscle pain and soreness on 10-point Likert scale
Overall muscular fatigue score | 5 days
  Subjective rating of overall muscular fatigue on a 12-cm visual analog scale

CONTACTS AND LOCATIONS:
Locations (1):
- VA Northern California Health Care System, Sacramento, California, United States

REFERENCES:
- [Derived] Hoffman MD, Badowski N, Chin J, Stuempfle KJ. A Randomized Controlled Trial of Massage and Pneumatic Compression for Ultramarathon Recovery. J Orthop Sports Phys Ther. 2016 May;46(5):320-6. doi: 10.2519/jospt.2016.6455. Epub 2016 Mar 23. PMID 27011305